CLINICAL TRIAL: NCT06047561
Title: The Scottish Aortic Stenosis LongiTudinal Imaging and biomarkeR (SALTIRE) Programme
Acronym: SALTIRE
Status: Recruiting | Type: Observational
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Other Study IDs: AC22131; RG/F/22/110093 (Other Grant/Funding Number: British Heart Foundation)
Record Dates: First submitted 2023-08-18; First posted 2023-09-21 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Aortic Stenosis
Keywords: Aortic Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Aortic Stenosis: Participants with Aortic Stenosis across the spectrum of disease severity
  Interventions: Radiation: PET-CT
- Aortic Valve Replacement: Participants who have previously undergone aortic valve replacement
  Interventions: Radiation: PET-CT
- Healthy Volunteers: Healthy Volunteers for the purposes of case-control analysis
  Interventions: Radiation: PET-CT

INTERVENTIONS:
Radiation: PET-CT — PET combined with CT or MRI
  Other Names: Positron Emission Tomography

SUMMARY:
The goal of this observational study is to understand the processes of what causes and accelerates the disease progress in aortic stenosis and following aortic valve replacement.

Participants will undergo transthoracic echocardiography every 6 months, with annual visits for state-of-the-art scanning techniques including positron-emission tomography combined with computed tomography or magnetic resonance imaging with radiotracers designed to look at disease processes including fibrosis, calcification, inflammation and thrombosis activity.

DETAILED DESCRIPTION:
This will be an observational cohort study using existing and prospectively recruited cohorts for both cross-sectional and longitudinal comparison across the spectrum of aortic stenosis severity. For existing cohorts of patients who have previously undergone research assessments, we will invite them for repeated assessments.

Participants will be reviewed every 6 months in the Clinical Research Facility (CRF) over a 4-year period. They will undergo clinical assessment, blood sampling, transthoracic echocardiography and advanced imaging annually including CT angiography, magnetic resonance and positron emission tomography (PET).

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged >50 years
* Provision of informed consent prior to any study specific procedures
* Patients with bioprosthetic aortic valve replacements, including both surgically and transcatheter implanted valves
* Patients with severe aortic stenosis (peak velocity >4.0 m/s; previously recruited patients)
* Patients with moderate aortic stenosis (peak velocity 3.0-4.0 m/s; new prospectively recruited patients)
* Patients with mild aortic stenosis (peak velocity 2.5-2.9 m/s; new prospectively recruited patients)
* Patients with aortic sclerosis (tri-leaflet thickened aortic valve with no obstruction of ventricular outflow)
* Age and sex-matched healthy volunteers

Exclusion Criteria:

* Inability or unwilling to give informed consent.
* Those with an allergy to iodinated contrast
* Patients with impaired renal function (eGFR of <30 mL/min/1.73m2)
* Women who are pregnant or breastfeeding.
* Patients with known Rheumatic Heart Disease
* Patients with known Ochronosis
* Patients with known Familial Homozygous Hypercholesterolaemia

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We will recruit up to 300 patients with aortic valve disease across the spectrum of disease severities from aortic sclerosis through to mild, moderate and severe aortic stenosis as defined by the European Society of Cardiology. We will also include those who have undergone bioprosthetic aortic valve replacement, and age and sex-matched control subjects with normal aortic valves.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-05-22 (Actual); Primary Completion 2028-05-22 (Estimated); Study Completion 2028-05-22 (Estimated)

PRIMARY OUTCOMES:
Haemodynamic aortic valve disease progression. | 4 years
  Rate of change of maximal aortic valve jet velocity (AV Vmax)

SECONDARY OUTCOMES:
Inflammatory, thrombotic, fibrotic and calcific aortic valve disease progression. | 4 years
  Rate of change of tissue-to-background ratio (TBRmax) of FDG, GP1, FAPI and NaF PET.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Edinburgh, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, CSR
Time Frame: End of Study to 15 years